CLINICAL TRIAL: NCT02331849
Title: Esophageal Motility in Eosinophilic Esophagitis Evaluated by High Resolution Manometry - Effect on Esophageal Motility of Standard Therapy.
Brief Title: Esophageal Motility in Eosinophilic Esophagitis Evaluated by High Resolution Manometry.
Acronym: HIMEOS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Technical University of Munich (Other)
Responsible Party: Principal Investigator, Monther Bajbouj, PD Dr. med., Technical University of Munich
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: HIMEOS-2013
Record Dates: First submitted 2013-12-02; First posted 2015-01-06 (Estimated); Last update posted 2015-01-06 (Estimated); Status verified 2015-01

CONDITIONS: Eosinophilic Esophagitis
Keywords: Eosinophilic esophagitis (EoE); GERD; esophageal motility
MeSH Terms: conditions — Eosinophilic Esophagitis; Gastroesophageal Reflux

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Eosinophilic esophagitis (Other): Patients with eosinophilic esophagitis after exclusion of GERD
  Interventions: Device: High resolution manometry (HRM)

INTERVENTIONS:
Device: High resolution manometry (HRM) — High resolution manometry of the esophagus

SUMMARY:
Esophageal Motility in eosinophilic esophagitis will be evaluated by High Resolution Manometry before and after medical treatment - motility is suspected to change/improve after therapy.

DETAILED DESCRIPTION:
After identification of eosinophilic inflammation of the esophagus -> differentiation between GERD and eosinophilic esophagitis (via pH/MII-measurements or PPI-trial) -> High-resolution manometry (HRM) for evaluation of esophageal motility in patients with eosinophilic esophagitis (exclusion of GERD-patients)-> initiation of budesonide-therapy -> after eight weeks of therapy reevaluation of esophageal motility by HRM

ELIGIBILITY:
Inclusion Criteria:

• patients with eosinophilic inflammation of the esophagus

Exclusion Criteria:

* refusal to participate in study
* pregnancy
* eosinophilic gastroenteritis
* Achalasia
* contraindication for gastroscopy / HRM / 24-h-pH/Impedance-monitoring
* contraindication for therapy with budesonide
* eosinophilic inflammation due to GERD

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2013-10; Primary Completion 2015-02 (Estimated)

PRIMARY OUTCOMES:
Improvement of esophageal motility (IBP) measureable in high resolution manometry (HRM) | Two months
  Average maximum intra-bolus-pressure (IBP) [mmHg] before and after therapy

SECONDARY OUTCOMES:
Improvement of esophageal motility (e.g. specified in the chicago classification) represented in high resolution manometry (HRM) | Two months
  weak peristalsis with small/large breaks, frequently failes peristalsis, absent peristalsis, hypertensive peristalsis, rapid contractions with normal latency, functional EGJ-obstruction, panesophageal pressurizations, compartimentalized pressurizations;
Endoscopic evaluation of inflammation before/after therapy | Two months
  Endoscopic assessment of esophageal signs of eosinophilic esophagitis (white exsudates, furrows, edema, rings, crepe paper, stricture
Symptoms before/after therapy | Two months
  Evaluation of symptoms via questionnaire before/after therapy

CONTACTS AND LOCATIONS:
Overall Officials: Simon Nennstiel, Dr. med., Principal Investigator — Klinikum rechts der Isar, II. Med. Klinik; Christoph Schlag, Dr. med., Principal Investigator — Klinikum rechts der Isar, II. Med. Klinik; Monther Bajbouj, PD Dr. med., Principal Investigator — Klinikum rechts der Isar, II. Med. Klinik
Locations (1):
- Klinikum rechts der Isar, II. Medizinische Klinik, München, Germany

REFERENCES:
- [Derived] Weidlich S, Nennstiel S, Jesinghaus M, Brockow K, Slotta-Huspenina J, Bajbouj M, Schmid RM, Schlag C. IgG4 is Elevated in Eosinophilic Esophagitis but Not in Gastroesophageal Reflux Disease Patients. J Clin Gastroenterol. 2020 Jan;54(1):43-49. doi: 10.1097/MCG.0000000000001154. PMID 30614939